CLINICAL TRIAL: NCT02062463
Title: A 12-Week, Randomized, Open-Label, Parallel-Group Study to Evaluate the Mastery of Inhaler Technique for Budesonide Formoterol (BF) SPIROMAX® (160/4.5 and 320/9 mcg) as Compared With SYMBICORT® TURBOHALER® (200/6 and 400/12 mcg) as Treatment for Adult Patients With Asthma (The Easy Low Instruction Over Time [ELIOT] Study)
Brief Title: Study to Evaluate the Mastery of Inhaler Technique for Budesonide Formoterol (BF) SPIROMAX® as Compared to SYMBICORT® TURBOHALER® as Treatment for Adult Participants With Asthma
Acronym: ELIOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFS-AS-40035; 2013-004630-14 (EudraCT Number)
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage 1: Empty Spiromax Followed by Empty Turbohaler (No Intervention): Participants will be trained on the proper use of empty Spiromax followed by empty Turbohaler devices.
- Stage 1: Empty Turbohaler Followed by Empty Spiromax (No Intervention): Participants will be trained on the proper use of empty Turbohaler followed by empty Spiromax devices.
- Stage 2: BF Spiromax (Experimental): Participants who have currently received 800 to 1000 micrograms (μg) beclomethasone-equivalent inhaled corticosteroid (ICS) per day will receive budesonide/formoterol twice daily using the BF Spiromax 160/4.5 device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax will be 640 μg and 18 μg, respectively. Participants who have currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day will receive budesonide/formoterol twice daily using the BF Spiromax 320/9 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax will be 1280 μg and 36 μg, respectively.
  Interventions: Drug: Budesonide and formoterol fumarate dehydrate (BF) SPIROMAX
- Stage 2: Symbicort Turbohaler (Active Comparator): Participants who have currently received 800 to 1000 μg beclomethasone-equivalent ICS per day will receive budesonide/formoterol twice daily using the Symbicort Turbohaler 200/6 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler will be 800 μg and 24 μg respectively. Participants who have currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day will receive budesonide/formoterol twice daily using the Symbicort Turbohaler 400/12 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler will be 1600 μg and 48 μg respectively.
  Interventions: Drug: SYMBICORT TURBOHALER budesonide and formoterol fumarate

INTERVENTIONS:
Drug: Budesonide and formoterol fumarate dehydrate (BF) SPIROMAX — SPIROMAX (BF) Budesonide and formoterol fumarate dehydrate (160/4.5 and 320/9 μg)
  Other Names: SPIROMAX®
  Arms: Stage 2: BF Spiromax
Drug: SYMBICORT TURBOHALER budesonide and formoterol fumarate — SYMBICORT® TURBOHALER® (200/6 and 400/12 μg)
  Other Names: SYMBICORT®; TURBOHALER®
  Arms: Stage 2: Symbicort Turbohaler

SUMMARY:
This study is conducted to assess whether training participants on proper use of BF SPIROMAX and Symbicort TURBOHALER will improve their device-handling technique and potentially improve their treatment outcome, that is, better asthma control.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of asthma in accordance with Global Initiative for Asthma (GINA) criteria as evidenced by a United Kingdom (UK) quality outcome framework approved Read code (UK diagnostic coding system).
* The participant is receiving step 3 or 4 therapy for asthma as defined by the British Thoracic Society (BTS) guidelines (daily doses of beclomethasone dipropionate [BDP]-equivalent ICS) ≥800 mcg to 2000 μg as part of fixed- or free combinations with long-acting β2-agonists (LABA).
* If participant is a female of childbearing potential (post-menarche or less than 2 years post-menopausal or not surgically sterile), the participant must be willing to commit to using a medically accepted method of contraception for the duration of study and 30 days after discontinuing study drug.
* The participant, as judged by the investigator, must be willing and able to understand risks and benefits of study participation to give informed consent and to comply with all study requirements as specified in this protocol for the entire duration of their study participation.
* The participant is SPIROMAX and TURBOHALER naïve (no use of a SYMBICORT TURBOHALER device in the last 6 months, minimizing carryover from prior device use).
* If female and of childbearing potential, the participant must have a negative urine pregnancy test.

  * other criteria apply, please contact the investigator for additional information.

Exclusion Criteria:

* The participant has any clinically significant uncontrolled medical condition (treated or untreated) that, in the judgment of the investigator, will cause participation in the study to be detrimental to the participant.
* The participant has participated in a Teva-sponsored clinical study with BF SPIROMAX in the last 6 months.
* The participant is a pregnant, attempting to become pregnant, or breast feeding. (Any woman becoming pregnant during the study will be withdrawn from the study.)
* The participant has used a clinical trial investigational drug within 1 month before the screening visit.
* The participant has an ongoing asthma exacerbation or has received OCS and/or antibiotics for a lower respiratory condition (proxy measure for identifying an asthma exacerbation and/or lower respiratory infection, suggestive of altered inspiratory capabilities) in the 2 weeks preceding visit 1.
* The participant is currently receiving any OCS (including long or short courses).
* The participant has a significant chronic lower respiratory tract disease other than asthma (for example chronic obstructive pulmonary disease [COPD], cystic fibrosis or interstitial lung disease). Conditions that are not predominant, such as minor degrees of bronchiectasis, are not a reason for exclusion.
* The participant has a known allergy or severe sensitivity to the constituents of the study drugs (SPIROMAX or TURBOHALER),for example, to lactose or to milk protein.

  * other criteria apply, please contact the investigator for additional information.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (74):
- United Kingdom (74):
  - Teva Investigational Site 34092, Axbridge
  - Teva Investigational Site 34081, Babbacombe
  - Teva Investigational Site 34103, Beccles
  - Teva Investigational Site 34144, Bishop's Stortford
  - Teva Investigational Site 34066, Burnhope
  - Teva Investigational Site 34064, Bury St Edmunds
  - Teva Investigational Site 34107, Bury St Edmunds
  - Teva Investigational Site 34072, Cheltenham
  - Teva Investigational Site 34063, Chippenham
  - Teva Investigational Site 34122, Chipping Norton
  - Teva Investigational Site 34134, Clacton-on-Sea
  - Teva Investigational Site 34136, Colchester
  - Teva Investigational Site 34143, Colchester
  - Teva Investigational Site 34111, Colchester
  - Teva Investigational Site 34126, Colchester
  - Teva Investigational Site 34135, Colchester
  - Teva Investigational Site 34120, Colchester
  - Teva Investigational Site 34075, Daventry
  - Teva Investigational Site 34112, Daventry
  - Teva Investigational Site 34083, East Hunsbury
  - Teva Investigational Site 34145, East Tillbury
  - Teva Investigational Site 34099, Exmouth
  - Teva Investigational Site 34110, Exmouth
  - Teva Investigational Site 34102, Goldhay
  - Teva Investigational Site 34119, Great Yarmouth
  - Teva Investigational Site 34079, Harrogate
  - Teva Investigational Site 34068, Harrogate
  - Teva Investigational Site 34139, Hemel Henpstead
  - Teva Investigational Site 34142, Hinckley
  - Teva Investigational Site 34116, Huntingdon
  - Teva Investigational Site 34113, Ipswich
  - Teva Investigational Site 34098, Lancashire
  - Teva Investigational Site 34128, Leicester
  - Teva Investigational Site 34127, Leicester
  - Teva Investigational Site 34141, Leigh-on-Sea
  - Teva Investigational Site 34082, Liskeard
  - Teva Investigational Site 34146, Lister House
  - Teva Investigational Site 34147, Liverpool
  - Teva Investigational Site 34080, Loughborough
  - Teva Investigational Site 34086, Lowestoft
  - Teva Investigational Site 34138, Luton
  - Teva Investigational Site 34076, Manchester
  - Teva Investigational Site 34109, Newton Aycliffe
  - Teva Investigational Site 34095, Norwich
  - Teva Investigational Site 34108, Norwich
  - Teva Investigational Site 34106, Norwich
  - Teva Investigational Site 34091, Norwich
  - Teva Investigational Site 34123, Norwich
  - Teva Investigational Site 34085, Oadby
  - Teva Investigational Site 34070, Oldham
  - Teva Investigational Site 34114, Orby
  - Teva Investigational Site 34118, Oxon
  - Teva Investigational Site 34137, Pickering
  - Teva Investigational Site 34124, Reading
  - Teva Investigational Site 34089, Redditch
  - Teva Investigational Site 34100, Sheringham
  - Teva Investigational Site 34117, Stalham
  - Teva Investigational Site 34105, Stanley
  - Teva Investigational Site 34065, Stowmarket
  - Teva Investigational Site 34067, Strensall
  - Teva Investigational Site 34078, Swindon
  - Teva Investigational Site 34140, Thaxted
  - Teva Investigational Site 34096, Thornton-Cleveleys
  - Teva Investigational Site 34088, Trowbridge
  - Teva Investigational Site 34077, Trowbridge
  - Teva Investigational Site 34071, Waterlooville
  - Teva Investigational Site 34073, Waterlooville
  - Teva Investigational Site 34084, Wells-Next-Sea
  - Teva Investigational Site 34115, Wisbech
  - Teva Investigational Site 34069, Woodbridge
  - Teva Investigational Site 34074, Woodbridge
  - Teva Investigational Site 34090, Worcester
  - Teva Investigational Site 34121, Wymondham
  - Teva Investigational Site 34101, York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in 2 stages: Stage 1 and 2. In Stage 1, participants were randomly assigned to either empty Spiromax followed by empty Turbohaler or empty Turbohaler followed by empty Spiromax. Stage 2 comprised randomization of eligible participants to the study drugs.
Groups:
- Stage 1: Empty Spiromax Followed by Empty Turbohaler: Participants were trained on the proper use of empty Spiromax followed by empty Turbohaler devices.
- Stage 1: Empty Turbohaler Followed by Empty Spiromax: Participants were trained on the proper use of empty Turbohaler followed by empty Spiromax devices.
- Stage 2: BF Spiromax: Participants who had currently received 800 to 1000 micrograms (μg) beclomethasone-equivalent inhaled corticosteroid (ICS) per day received budesonide/formoterol twice daily using the BF Spiromax 160/4.5 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 640 μg and 18 μg, respectively. Participants who had currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the BF Spiromax 320/9 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 1280 μg and 36 μg, respectively.
- Stage 2: Symbicort Turbohaler: Participants who had currently received 800 to 1000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 200/6 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 800 μg and 24 μg respectively. Participants who had currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 400/12 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 1600 μg and 48 μg respectively.
Period: Crossover Stage 1
Arm/Group | Stage 1: Empty Spiromax Followed by Empty Turbohaler | Stage 1: Empty Turbohaler Followed by Empty Spiromax | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Started | 243 | 242 | 0 | 0
Full Analysis Set (All randomized participants who completed assessments on both study devices (empty Turbohaler and empty Spiromax), permitting a paired analysis of results.) | 240 | 241 | 0 | 0
Completed | 240 | 241 | 0 | 0
Not Completed | 3 | 1 | 0 | 0
Not completed — Withdrawals during stage 1 were not captured | 3 | 1 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: Empty Spiromax Followed by Empty Turbohaler | Stage 1: Empty Turbohaler Followed by Empty Spiromax | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Started | 0 | 0 | 197 | 197
Received at Least 1 Dose of Study Drug | 0 | 0 | 197 | 197
Full Analysis Set (All randomized participants who returned for assessment of maintenance of inhaler technique at Week 12, and who had at least 10 weeks (inclusive) of device use of the inhaler (treatment) to which they were randomly assigned.) | 0 | 0 | 151 | 154
Completed | 0 | 0 | 144 | 141
Not Completed | 0 | 0 | 53 | 56
Not completed — Adverse Event | 0 | 0 | 12 | 20
Not completed — Lack of Efficacy | 0 | 0 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 20 | 20
Not completed — Non-Compliance | 0 | 0 | 0 | 1
Not completed — Other than specified | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 15 | 10

BASELINE CHARACTERISTICS:
Population: Randomized analysis set included all randomized participants.
Groups:
- Empty Spiromax Followed by Empty Turbohaler: Participants were trained on the proper use of empty Spiromax followed by empty Turbohaler devices.
- Empty Turbohaler Followed by Empty Spiromax: Participants were trained on the proper use of empty Turbohaler followed by empty Spiromax devices.
- Total: Total of all reporting groups
Arm/Group | Empty Spiromax Followed by Empty Turbohaler | Empty Turbohaler Followed by Empty Spiromax | Total
Number analyzed (Participants) | 243 | 242 | 485
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.8) | 53.1 (14.2) | 53.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 134 | 286
  Male | 91 | 108 | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 238 | 235 | 473
  Black | 1 | 2 | 3
  Asian | 3 | 3 | 6
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants Achieving Device Mastery
Description: Device mastery was defined as absence of healthcare professional (HCP)-observed errors by the end of Step 3 of a 6-step standardized device training protocol for empty Spiromax compared to empty Turbohaler. The 6 steps of device training protocol were: Step 1 - Intuitive use; Step 2 - Patient information leaflet; Step 3 - Instructional video; Step 4 - HCP tuition; Step 5 - HCP tuition (1st repeat); Step 6 - HCP tuition (2nd repeat).
Time Frame: Baseline (Day 1)
Population: Full analysis set (FAS) for Stage 1 included all randomized participants who completed assessments on both study devices (empty Turbohaler and empty Spiromax), permitting a paired analysis of results.
Measure: Number; unit: percentage of participants
Groups:
- Stage 1: Empty Spiromax: Participants were trained on the proper use of empty Spiromax.
- Stage 1: Empty Turbohaler: Participants were trained on the proper use of empty Turbohaler.
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 481 | 481
percentage of participants | 94.4 | 86.9
Statistical Analysis 1: Comparison: Stage 1: Empty Spiromax vs Stage 1: Empty Turbohaler; Analysis was performed using a conditional logistic regression model; Test type: Other; p < 0.001, Chi-squared — Threshold for significance at 0.05 level; Odds Ratio (OR) = 3.77, 95% CI 2-sided [2.05 to 6.95]

2. Primary Outcome: Stage 2: Percentage of Participants Maintaining Device Mastery
Description: Maintenance of device mastery was defined as absence of HCP-observed errors after 12 weeks of device use.
Time Frame: Baseline up to Week 12
Population: FAS for Stage 2 included all randomized participants who returned for assessment of maintenance of inhaler technique at Week 12, and who had at least 10 weeks (inclusive) of device use of the inhaler (treatment) to which they were randomly assigned.
Measure: Number; unit: percentage of participants
Groups:
- Stage 2: BF Spiromax: Participants who had currently received 800 to 1000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the BF Spiromax 160/4.5 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 640 μg and 18 μg, respectively. Participants who had currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the BF Spiromax 320/9 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 1280 μg and 36 μg, respectively.
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
percentage of participants | 58.9 | 53.2
Statistical Analysis 1: Comparison: Stage 2: BF Spiromax vs Stage 2: Symbicort Turbohaler; Analysis was performed using a conditional logistic regression model; Test type: Other; p = 0.316, Chi-squared — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.80 to 1.98]

3. Secondary Outcome: Stage 1: Percentage of Participants Achieving Device Mastery by Step 1
Description: The number of participants achieving device mastery by Step 1 (no training/intuitive use) of the device training process. Device mastery was defined as the absence of nurse-observed errors by the end of Step 3 of a 6-step standardized device training protocol for each device. The 6 training steps were as follows: Step 1, intuitive use; Step 2, patient device information leaflet; Step 3, instructional video; Step 4, nurse tuition; Step 5, nurse tuition (1st repeat); Step 6, nurse tuition (2nd repeat). After each training step an assessment of device use was carried out by the nurse using a pre-defined list of inhaler errors.
Time Frame: Day 1
Population: FAS for Stage 1 included all randomized participants who completed assessments on both study devices (empty Turbohaler and empty Spiromax), permitting a paired analysis of results.
Measure: Number; unit: Percentage of participants
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 481 | 481
Percentage of participants | 33.3 | 11.4

4. Secondary Outcome: Stage 1: Percentage of Participants Achieving Device Mastery by Step 2
Description: The number of participants achieving device mastery by Step 2 (patient device information leaflet) of the device training process. Device mastery was defined as the absence of nurse-observed errors by the end of Step 3 of a 6-step standardized device training protocol for each device. The 6 training steps were as follows: Step 1, intuitive use; Step 2, patient device information leaflet; Step 3, instructional video; Step 4, nurse tuition; Step 5, nurse tuition (1st repeat); Step 6, nurse tuition (2nd repeat). After each training step an assessment of device use was carried out by the nurse using a pre-defined list of inhaler errors.
Time Frame: Day 1
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 481 | 481
Percentage of participants | 80.2 | 64.0

5. Secondary Outcome: Stage 1: Number of Steps Taken to Achieve Device Mastery
Time Frame: Baseline (Day 1)
Population: as for outcome 3
Measure: Median (Full Range); unit: steps
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 481 | 481
steps | 1 [0 to 12] | 2 [0 to 15]

6. Secondary Outcome: Stage 1: Number of Nurse-Observed Errors
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 481 | 481
Errors | 1.91 (0.89) | 2.36 (0.92)

7. Secondary Outcome: Stage 1: Patient Satisfaction and Preference Questionnaire (PASAPQ) Total Score
Description: The PASAPQ is a multi-item measure of inhalation device satisfaction and preference designed specifically for participants with asthma and chronic obstructive pulmonary disease. The PASAPQ includes a total of 14 device satisfaction items, including an overall satisfaction item. The total score was the sum of the 13 items related to performance and convenience domains (7 items for performance domain: Questions 1-5, 10-11, and 6 items for convenience domain: Questions 6-9, 12-13). Each PASAPQ item had response options ranging from 1 (very dissatisfied) to 7 (very satisfied). To calculate the total score, the items within each domain were first summed and then transformed to a 0 (least) or 100 (most) point scale, with higher scores indicating greater satisfaction.
Time Frame: Baseline (Day 1)
Population: FAS for Stage 1 included all randomized participants who completed assessments on both study devices (empty Turbohaler and empty Spiromax), permitting a paired analysis of results. Here 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Stage 1: Empty Spiromax | Stage 1: Empty Turbohaler
Number analyzed (Participants) | 477 | 477
units on a scale | 89.80 [18.37 to 100.00] | 85.71 [14.29 to 100.00]

8. Secondary Outcome: Composite Endpoint: Stage 2: Total Number of Observed Errors (Nurse and Technology [Vitalograph Pneumotrac Spirometer])
Description: Composite score calculated as the sum of nurse observed errors and technology-observed errors.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
errors | 0.50 (0.68) | 0.82 (1.10)

9. Secondary Outcome: Stage 2: Number of Technology-Observed Errors (Vitalograph Pneumotrac Spirometer)
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Errors
Groups:
- Stage 1: Symbicort Turbohaler: Participants who had currently received 800 to 1000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 200/6 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 800 μg and 24 μg respectively. Participants who had currently received 1600 to 2000 μg beclomethasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 400/12 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 1600 μg and 48 μg respectively.
Arm/Group | Stage 2: BF Spiromax | Stage 1: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
Errors | 0.01 (0.08) | 0.01 (0.08)

10. Secondary Outcome: Stage 2: Total Number of Handling Errors
Description: Total number of device handling errors included HCP observed errors and technology observed errors.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
errors | 0.50 (0.68) | 0.82 (1.10)

11. Secondary Outcome: Stage 2: Change in Handling Errors From Stage 1 to Stage 2
Description: The difference in the number of handling errors identified after participant training using the patient device information leaflet at stage 1 and after 12 weeks of treatment (end of stage 2).
Time Frame: Baseline (Day 1), Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Errors
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
Errors | -0.95 (1.72) | -2.01 (2.52)

12. Secondary Outcome: Stage 2: Number of Participants In Pre-specified Treatment Adherence Categories (Assessed by Device Dose Counters)
Description: Treatment adherence was categorized (as less than or equal to 50%, 51%-70%, 71%-99%, and 100%) and compared across treatment groups using a chi-square test.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
Participants
  ≤50% | 60 | 61
  51-70% | 19 | 16
  71-99% | 70 | 71
  100% | 2 | 6

13. Secondary Outcome: Stage 2: Change From Baseline in 6-Item Asthma Control Questionnaire (ACQ) (Excluding Forced Expiratory Volume in 1 Second [FEV1] Question) Score at Weeks 4, 8, and 12
Description: The ACQ is a 7-item, validated tool for assessing asthma control (Juniper et al 1999). Thinking about their asthma for the last 7 days, participants were asked to evaluate their asthma against 5 symptom items and a rescue bronchodilator use question using a 7-point scale (0=no impairment and 6=maximum impairment). Spirometry data were used to grade the percent predicted forced expiratory volume in 1 second (FEV1) on a 7-point scale (0 to 6). The score is the mean of the first 6 questions (excluding the FEV1 question), generating a value from 0 (totally controlled) to 6 (severely uncontrolled). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Weeks 4, 8, and 12
Population: FAS for Stage 2 included all randomized participants who returned for assessment of maintenance of inhaler technique at Week 12, and who had at least 10 weeks (inclusive) of device use of the inhaler (treatment) to which they were randomly assigned. Here 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 142 | 147
units on a scale
  Change at Week 4: number analyzed (Participants) | 142 | 140
  Change at Week 4 | -0.22 (0.83) | -0.33 (0.81)
  Change at Week 8: number analyzed (Participants) | 140 | 143
  Change at Week 8 | -0.20 (0.98) | -0.30 (1.04)
  Change at Week 12: number analyzed (Participants) | 137 | 147
  Change at Week 12 | -0.22 (0.95) | -0.36 (1.05)

14. Secondary Outcome: Stage 2: Change From Baseline in 7-Item ACQ
Description: The ACQ is a 7-item, validated tool for assessing asthma control (Juniper et al 1999). Thinking about their asthma for the last 7 days, participants were asked to evaluate their asthma against 5 symptom items and a rescue bronchodilator use question using a 7-point scale (0=no impairment and 6=maximum impairment). Spirometry data were used to grade the percent predicted FEV1 on a 7-point scale (0 to 6). The ACQ score is the mean of the 7 questions, generating a value from 0 (totally controlled) to 6 (severely uncontrolled). A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 145 | 149
units on a scale | -0.20 (0.78) | -0.31 (0.92)

15. Secondary Outcome: Stage 2: Time to First Treatment Failure
Description: Time to treatment failure was defined as change of asthma treatment or treatment for an asthma exacerbation or lower respiratory tract infection.
Time Frame: Baseline up to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
days | 76.38 (21.42) | 73.95 (24.27)

16. Secondary Outcome: Stage 2: Number of Participants With Severe Asthma Exacerbations
Description: Severe asthma exacerbation was defined as a hospitalization or emergency room attendance for asthma, or an acute course of oral corticosteroids (OCS).
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
Participants
  0 asthma exacerbation | 139 | 136
  1 asthma exacerbation | 11 | 17
  2 asthma exacerbation | 1 | 1
  ≥3 asthma exacerbations | 0 | 0

17. Secondary Outcome: Stage 2: Impact of Maintaining Device Mastery on Time to Treatment Failure
Description: The impact of maintaining device mastery on time to treatment failure (defined as change of asthma treatment or treatment for an asthma exacerbation or lower respiratory tract infection) was assessed by comparing the time to treatment failure for participants with and without device mastery. Device mastery was defined as the absence of nurse-observed errors by the end of Step 3 of a 6-step standardized device training protocol for each device.
Time Frame: Baseline Up to Week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Stage 2: BF Spiromax | Stage 1: Symbicort Turbohaler
Number analyzed (Participants) | 151 | 154
Days
  Device mastery = Yes: number analyzed (Participants) | 89 | 82
  Device mastery = Yes | 72.99 (22.38) | 75.93 (22.59)
  Device mastery = No: number analyzed (Participants) | 62 | 72
  Device mastery = No | 81.24 (19.11) | 71.69 (26.03)

18. Secondary Outcome: Stage 2: Impact of Maintaining Device Mastery on Asthma Control Questionnaire Score
Description: The impact of maintaining device mastery on asthma control was assessed by comparing the 7-item ACQ scores for participants with and without device mastery. The ACQ is a 7-item, validated tool for assessing asthma control (Juniper et al 1999). Thinking about their asthma for the last 7 days, participants were asked to evaluate their asthma against 5 symptom items and a rescue bronchodilator use question using a 7-point scale (0=no impairment and 6=maximum impairment). Spirometry data were used to grade the percent predicted FEV1 on a 7-point scale (0 to 6). The ACQ score is the mean of the 7 questions, generating a value from 0 (totally controlled) to 6 (severely uncontrolled). Device mastery was defined as the absence of nurse-observed errors by the end of Step 3 of a 6-step standardized device training protocol for each device.
Time Frame: Baseline Up to Week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 145 | 149
Units on a scale
  Device mastery = Yes: number analyzed (Participants) | 85 | 79
  Device mastery = Yes | 1.25 (1.05) | 1.35 (0.95)
  Device mastery = No: number analyzed (Participants) | 60 | 70
  Device mastery = No | 1.46 (0.97) | 1.37 (0.97)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to Week 12
Population: The safety population for stage 2 included all participants randomly assigned to treatment who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
Number analyzed (Participants) | 197 | 197
Participants | 113 | 119

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Per planned analysis no adverse events were collected or reported during Stage 1.
  For the purpose of adverse event recording, the study period was defined for each participant as the time period from randomization of treatment in stage 2 through the end of the treatment period.
  The safety population for stage 2 included all participants randomly assigned to treatment who received at least 1 dose of study drug.
Groups:
- Stage 2: BF Spiromax: Participants who had currently received 800 to 1000 μg beclometasone-equivalent ICS per day received budesonide/formoterol twice daily using the BF Spiromax 160/4.5 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 640 μg and 18 μg, respectively. Participants who had currently received 1600 to 2000 μg beclometasone-equivalent ICS per day received budesonide/formoterol twice daily using the BF Spiromax 320/9 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using BF Spiromax were 1280 μg and 36 μg, respectively.
- Stage 2: Symbicort Turbohaler: Participants who had currently received 800 to 1000 μg beclometasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 200/6 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 800 μg and 24 μg respectively. Participants who had currently received 1600 to 2000 μg beclometasone-equivalent ICS per day received budesonide/formoterol twice daily using the Symbicort Turbohaler 400/12 μg device. Therefore, the daily, ex-mouthpiece doses of budesonide and formoterol using Symbicort Turbohaler were 1600 μg and 48 μg respectively.
Arm/Group | Stage 2: BF Spiromax | Stage 2: Symbicort Turbohaler
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/197
Serious Adverse Events (participants affected / at risk) | 3/197 | 7/197
Other Adverse Events (participants affected / at risk) | 27/197 | 39/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2: BF Spiromax (N=197) | Stage 2: Symbicort Turbohaler (N=197)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2: BF Spiromax (N=197) | Stage 2: Symbicort Turbohaler (N=197)
Lower respiratory tract infection (Infections and infestations) | 16 (16) | 29 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.